CLINICAL TRIAL: NCT04772482
Title: Testing of Alternatives for Dark Hair Dyes in Patients With Proven Sensitization to Para-Phenylenediamine
Brief Title: Study on Hypoallergenic Hair Dye
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: DERM-2020-29233
Record Dates: First submitted 2021-02-23; First posted 2021-02-26 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Contact Dermatitis; Allergy; Dermatitis; Dermatitis
MeSH Terms: conditions — Dermatitis, Contact; Dermatitis, Atopic; Dermatitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All Participants: All participants will undergo path testing to determine skin sensitivity to certain compounds.
  Interventions: Diagnostic Test: Sensitivity Patch Testing

INTERVENTIONS:
Diagnostic Test: Sensitivity Patch Testing — Testing patches will be applied on the upper arms. Para-phenylene diamine (PPD) 1% will be applied on one upper arm. Para-toluenediamine sulfate (PTD), 2-methoxyethyl p-phenylenediamine (ME-PPD), PPD6 and PPD7 will be applied to the other upper arm.

SUMMARY:
Permanent hair dyes are commonly used in over the counter direct to consumer products and within hair salons. Allergy, also known as contact dermatitis, to hair dye is a well known phenomenon. Herein, we seek to decrease the risks of allergy to hair dyes by testing a novel version of p-phenylenediamine (PPD) with less allergy potential.

DETAILED DESCRIPTION:
For patients with PPD sensitizations, it is important to find alternatives for dark hair dyes. P-toluenediamine (PTD) and potentially also 2-methoxyethyl p-phenylenediamine (ME-PPD) show cross-reactivity with PPD and therefore we want to prove that our new compounds PPD-6 and PPD-7 show no or significantly reduced cross-reactions with PPD and do not induce relevant allergic reactions in patients with proven PPD sensitizations.

Our specific aims for this study are the following:

A1) To show that PPD 6 and PPD 7 have reduced or optimally no reaction in standard patch tests in patients with proven allergy to PPD A2) To compare the sensitization pattern to other possible commercially available alternatives for hair dye, such as ME-PPD and PTD A3) To evaluate and rule out any possible non-specific irritant reaction of PPD-6 and PPD-7 in these patch tests (i.e. confirm in-vitro safety profile in-vivo)

ELIGIBILITY:
Inclusion Criteria:

- Proven Diagnosis of PPD and/or PTD sensitization (patch tests and clinically relevant eczematous reactions to hair dye)

Exclusion Criteria:

* Use of oral immunosuppressive, anti-inflammatory and chemotherapy medications, particularly corticosteroids for at least 1 month before testing.
* Immunocompromised patient (e.g. Cancer, Diabetes mellitus, medication, Immunodeficiency, radiation therapy)
* History of acute hepatitis, chronic liver disease or end stage liver disease.
* History of human immunodeficiency virus (HIV) or acquired immune deficiency syndrome.
* Use of illicit drugs within the past 6 months prior to study start and/or opioid use disorder.
* Pregnancy as established by questionnaire

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with sensitivity to PPD and/or PTD
Sampling Method: Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-05-13 (Actual); Study Completion 2022-05-13 (Actual)

PRIMARY OUTCOMES:
Allergy to Study Compounds | 4 days
  The primary endpoint of the study is the percent of participants with a known PPD allergy who experience an allergic reaction to the study compounds PPD6 or PPD7.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Bigliardi, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States